CLINICAL TRIAL: NCT00229580
Title: Health Behavior Feedback Study for Veterans With Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Alcoholic Beverage Medical Research Foundation (Other)
Responsible Party: Tania Correale, Ph.D., VA PSHCS/UWashington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-8752-V 03
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Alcoholism; Alcohol Abuse; Hepatitis C; Liver Disease
Keywords: Brief Intervention; Motivational Interviewing; Health Psychology; Alcohol; Hepatitis C; Patient Education
MeSH Terms: conditions — Alcoholism; Hepatitis C; Liver Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Motivational feedback
  Interventions: Behavioral: 3 session brief intervention with health behavior feedback
- 2 (Active Comparator): treatment as usual
  Interventions: Other: treatment as usual

INTERVENTIONS:
Behavioral: 3 session brief intervention with health behavior feedback
  Arms: 1
Other: treatment as usual
  Arms: 2

SUMMARY:
The purpose of this study was to explore whether a brief (3 session) intervention would impact health behavior of veterans with hepatitis C. The main focus of the intervention was on reduction of heavy drinking with patients who have liver disease. Other study goals were to increase the likelihood that patients would seek out substance use treatment and/or hepatitis C health care services. The study also tested the use of a liver function test called CDT/GGT in detecting heavy drinking. The main hypothesis was that a 3 session intervention with personalized feedback about health behavior would result in a reduction in alcohol use and increased use of substance use treatment and hepatology health care.

DETAILED DESCRIPTION:
OBJECTIVES: To establish the feasibility of a brief intervention for hepatitis C+ (HCV) patients who drink alcohol. The primary aim was reduction in alcohol use, which is known to be hazardous for patients with chronic HCV infection. Secondary aims were: 1) to increase patient engagement in substance use disorder (SUD) treatment, 2) to explore patient engagement in HCV specialty care, treatment acceptability, and impact on other health-related behaviors, and 3) to examine pre-post intervention differences in relation to report of alcohol use and to explore whether the CDT/GGT merits tracking to detect heavy drinking in this population, given hepatic pathology.

DESIGN: Randomized controlled trial with six-week and 12-week post-baseline assessment follow-up. The control group was offered the brief intervention at completion of the 12-week post-baseline follow-up.

PARTICIPANTS: We had anticipated recruiting 60 veterans who were HCV+, referred for HCV specialty care (education or treatment evaluation), and who met criteria for hazardous alcohol use. Due to problems with recruitment, only 12 veterans participated in the study (see below).

RECRUITMENT: We started regular study recruitment September 27, 2004 but study recruitment was much slower than anticipated. Despite multiple modifications to change our recruitment eligibility criteria, we enrolled only twelve subjects (N=12). Due to this ongoing recruitment problem, we decided to end study enrollment on 9/30/05 with follow-up completion in December 2005. Despite an extension of the Alcoholic Beverage Medical Research Foundation grant, there was no progress in identifying an alternative recruitment or developing an appropriate follow-up study.

MEASURES: Baseline assessment included demographic information, the Alcohol Use Disorders Identification Test (AUDIT), Form - 90 (recent alcohol and drug use), a DSM-IV SUD criteria checklist, a Health Behavior Questionnaire, and the K-10 (brief measure of psychological distress). For brief intervention feedback, the Short Inventory of Problems (negative consequences of alcohol use), the SOCRATES (stage of readiness to change), blood draw for liver function tests, and two brief measures of neuropsychological functioning were administered. VA treatment utilization data (SUD and specialty HCV treatment attendance) was obtained. Follow-up sessions also included measures of treatment acceptability and concept retention.

INTERVENTION: Participants in the brief intervention condition received personalized feedback and encouragement to explore ambivalence about change and treatment in three sessions. Feedback and interventions were tailored to individuals' health-related behavior with emphasis on alcohol use.

COMPLETION DATA: Ten participants were randomized to receive the feedback session and two were randomized to receive the treatment as usual or control group. Of the twelve participants enrolled, eight individuals (7 randomized, 1 control) completed all study sessions, one completed 2 of the 3 required sessions (1 control), and three who received the intervention completed only the initial baseline session.

DEMOGRAPHICS: We had eleven men and one female enroll in the study. The mean age of our participants was 55 years old. Five subjects identified themselves as African American or Black while seven identified themselves as Caucasian or White. Half (N=6) of the group were divorced and 42% (N=5) of the group were unemployed at the time they enrolled in the study. Over half (58%) of the subjects had completed some college in their lifetime.

SUD INFORMATION AND FEEDBACK: All subjects receiving the feedback sessions received a Personal Feedback Report at their first intervention session. This report incorporated data from the SOCRATES, SUD criteria checklist, Form 90 - revised, the SIP, and the Health Behavior Questionnaire which was collected at an earlier baseline session. For those receiving the feedback sessions (N=10), all had a primary diagnosis of alcohol dependence, while eight also endorsed use of additional substances (cocaine, opiates, cannabis and/or amphetamines).

Compared to individuals of the same gender in the population, the mean percentile rank of drinking norms was 97.5 (sd = 3.26). Based on data from the Form- 90 regarding typical weekly drinking patterns and levels of intoxication, the subjects in the feedback session had a reported mean Blood Alcohol Concentration (BAC) level of .13 (sd =.13) in a typical week, with a mean typical heavy day of drinking reaching a BAC of .23 (sd = .30). Subjects received feedback on the common effects of different levels of intoxication and how their self-reported drinking compared.

Besides receiving feedback on their drinking and the associated negative consequences, subjects also received feedback on their reported drug use. Cocaine and cannabis were the most frequently used drugs within the 30 days prior to the baseline, with subjects reporting mean use of 3.4 (sd = 6.7, sd =6.3, respectively) days out of 30. Subjects also received feedback on their smoking habits. Of the ten non-randomized subjects nine reported some tobacco use at baseline and no one reported decreased or discontinued use of tobacco after receiving the intervention.

TREATMENT ACCEPTABILITY: After the follow-up appointments we asked subjects (N=7) to rate their acceptance of the study intervention sessions on 14 different items ranging from their feelings of the discussions sessions to ratings on the therapist they met with throughout the study. Items were scored on a scale of 1-7. At the final follow-up 71% (N=5) reported the sessions as being valuable and easy to complete. Ninety percent (N=6) of the subjects who completed follow-up also reported the therapist as being helpful and caring towards them in the sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Positive serology for current infection by hepatitis C viremia by PCR confirmation test;
2. Current alcohol use (past 30 days) as indicated by self-report (using AUDIT- C questions);
3. Meets hazardous alcohol use criteria as measured by the Alcohol Use Disorders Identification Test.

   Criteria per (National Institute on Alcohol Abuse and Alcoholism, 1995):
   1. for women, 7 or more drinks per week or 4 or more drinks per occasion;
   2. for men, 14 or more drinks per week or 5 or more drinks per occasion;
4. Not currently engaged (past 30 days) in VA specialty substance use disorder treatment or mutual help groups like AA/NA.

Exclusion Criteria:

1. Abstinent from alcohol use in last 30 days as indicated by self-report or less than hazardous use according to criteria listed above by the AUDIT.
2. Patient is already engaged (past 30 days) in specialty substance use disorder treatment or attends self-help groups.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-12; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Reduction in alcohol consumption | at 6 and 12-week follow-up.

SECONDARY OUTCOMES:
Engagement in substance use treatment and hepatitis C specialty care. Detection of elevated CDT in blood serum compared with self-reported heavy drinking. | 12 weeks post-study

CONTACTS AND LOCATIONS:
Overall Officials: Tania M Davis Correale, PhD, Principal Investigator — Department of Psychiatry and Behavioral Sciences, University of Washington School of Medicine
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States